CLINICAL TRIAL: NCT03524417
Title: Effect of Equine Rabies Immunoglobulin Injection on Day 7 After First Dose of Rabies Vaccination to Rabies Immune Response
Brief Title: Effect of ERIG Injection on Day 7 After First Dose of Rabies Vaccination to Rabies Immune Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal investigator, Queen Saovabha Memorial Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2/2017
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Rabies
Keywords: Rabies immunoglobulin
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIG injection (Experimental): RIG injection on day 7
  Interventions: Biological: Equine rabies immunoglobulin injection on day 7

INTERVENTIONS:
Biological: Equine rabies immunoglobulin injection on day 7 — The patients with WHO category III rabies exposure, who have received first dose of rabies vaccination a week before and have not received rabies immunoglobulin were enrolled. Blood for Rabies neutralizing antibody titers (RNab) would be examined on day 0. On the same day, Equine rabies immunoglobulin (ERIG) at the dosage of 40 IU/kg would be injected into and around the wound as much as possible and the rest would be injected intramuscularly at the site distance from rabies vaccine. Then blood for RNab would be serially examined on day 7, 14, 90, 365.

SUMMARY:
No study was conducted to evaluate the rabies neutralizing antibody titers after RIG injection on day 7. The only study that has supported the delay of RIG administration was done in 1996 by our institute, of which RIG was given on day 5 with the original Thai Red Cross intradermal regimen (2-2-2-0-1-1).

DETAILED DESCRIPTION:
Rabies immunoglobulin (RIG) should be administered as soon as possible after the initiation of post-exposure prophylaxis. RIG should not be given after day 7 following the first rabies vaccine dose, because circulating neutralizing antibody will have begun to appear. Nevertheless, no study was conducted to evaluate the rabies neutralizing antibody titers after RIG injection on day 7.

The only study that has supported the delay of RIG administration was done in 1996 by our institute, of which RIG was given on day 5 with the original Thai Red Cross intradermal regimen (2-2-2-0-1-1). The ongoing study would prove the validity of the recommendation and eliminate the controversies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* WHO category III rabies exposure
* Received rabies vaccination on day 0 and 3.

Exclusion Criteria:

* Received RIG
* Immunocompromised hosts or receiving immunosuppressive therapy
* Received blood or blood product within 3 months
* Received anti-malarial drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rabies neutralizing antibody titers | Change from baseline of geometric mean titres of rabies neutralizing antibody titres at 2 weeks
  Rabies neutralizing antibody titers would be represented and compared by geometric mean titers (GMTs)

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Thai Red Cross Society, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided